CLINICAL TRIAL: NCT03461510
Title: Dysglycemia & Obesity: Impact on the Brain in Adolescents With Type 2 Diabetes
Brief Title: Type 2 Diabetes and the Brain in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Lydia Snyder, MD, Nemours Children's Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-35
Record Dates: First submitted 2018-01-04; First posted 2018-03-12 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Pediatric Obesity; Insulin Resistance; Dysglycemia; Hyperglycemia
Keywords: Cognition; MRI; Functional MRI; Pediatric Obesity; Type 2 Diabetes Mellitus; Adolescents; Continuous Glucose Monitoring; Insulin Clamp
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Pediatric Obesity; Insulin Resistance; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Type 2 Diabetes (Experimental): Hyperglycemic clamp and Hyperinsulinemic Euglycemic clamp
  Interventions: Procedure: Hyperglycemic clamp; Procedure: Hyperinsulinemic Euglycemic clamp
- Lean Control (No Intervention): Controls do not undergo Hyperglycemic clamp and Hyperinsulinemic Euglycemic clamp
- Obese Control (No Intervention): Controls do not undergo Hyperglycemic clamp and Hyperinsulinemic Euglycemic clamp

INTERVENTIONS:
Procedure: Hyperglycemic clamp — Subjects with T2D will receive IV Dextrose infusion to maintain plasma glucose at ~250 mg/dL during fMRI.
  Arms: Type 2 Diabetes
Procedure: Hyperinsulinemic Euglycemic clamp — Subjects with T2D will receive IV Dextrose and Insulin infusion to maintain plasma glucose at approximately 90 mg/dL during fMRI.
  Arms: Type 2 Diabetes

SUMMARY:
This study evaluates differences in brain function and cognitive performance in adolescents with type 2 diabetes (T2D) compared to non diabetic controls (both obese and lean) and correlates these changes with obesity, insulin resistance, and glycemic control in youth with T2D.

DETAILED DESCRIPTION:
This is a cross-sectional study examining neurocognitive function and brain activity in resting state and during working memory and executive function tasks using blood oxygen level dependent (BOLD) functional MRI (fMRI) during hyperinsulinemic euglycemic and hyperglycemic clamps in obese adolescents with T2D compared to non-diabetic obese and lean controls. The investigators will measure glycemic control (acute hyperglycemia during clamps and glycemic variability) and insulin resistance to examine their association with neurocognitive metrics and brain functional activity.

There will be one screening visit and three study visits for subjects with T2D. One visit will consist of neurocognitive testing and dual energy X-ray absorptiometry (DEXA) of the whole body to assess body composition including fat mass. In the other two visits, subjects with T2D will undergo normal and high glucose clamps during fMRI.

Obese and lean control subjects will have one screening visit and two study visits, one for neurocognitive testing and DEXA and another for fMRI without glucose clamps. All subjects will have a blood sample obtained at the screening visit.

Only adolescents with type 2 diabetes will wear a continuous glucose monitor (CGM) for 6 days prior to neuroimaging to determine glycemic variability. A1C will be assessed at baseline.

Parents of subjects will also have abbreviated IQ testing.

ELIGIBILITY:
Inclusion Criteria:

Type 2 Diabetes:

* BMI ≥85th percentile
* A1c ≥ 8%
* Pubertal

Healthy Controls:

* BMI ≥85th percentile for Obese Controls
* BMI < 85th percentile for Lean Controls
* Pubertal
* Normal A1c & Fasting glucose

Exclusion Criteria:

* Significant developmental delay or learning disability
* Significant visual or auditory deficits
* Born <34 weeks gestation
* Neurologic disease
* Psychiatric disease requiring inpatient treatment
* Significant head trauma
* Malignancy
* Pregnancy
* Weight > 350lb (MRI weight limit)
* Metal in the body (including dental braces)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Brain Activity using functional MRI (fMRI) | Baseline
  The investigators will examine functional connectivity of brain networks during cross sectional resting-state and task-related (working memory and response inhibition) BOLD-fMRI activation. fMRI activation in adolescents with T2D will be compared to age- and sex- matched, non-diabetic, healthy lean and obese controls.
Neurocognitive battery metrics including IQ as well as executive function and visual-spatial memory | Baseline
  The investigators will evaluate cognitive performance by examining test scores from neurocognitive metrics which reflect global IQ, spatial recognition, episodic memory, executive function (includes response inhibition, working memory), academic achievement, and processing speed. Adolescents with T2D will be compared to controls to determine whether these differences are associated with glycemic control, obesity, and insulin resistance.
fMRI performance in relation to dysglycemia | Baseline
  In adolescents with T2D, the investigators will examine BOLD-fMRI brain activation in relation to acute hyperglycemia during glucose clamping, chronic hyperglycemia, glycemic variability, and insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Snyder, MD, Principal Investigator — Nemours Children's Health System
Locations (1):
- Nemours Children's Health System, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mazaika PK, Weinzimer SA, Mauras N, Buckingham B, White NH, Tsalikian E, Hershey T, Cato A, Aye T, Fox L, Wilson DM, Tansey MJ, Tamborlane W, Peng D, Raman M, Marzelli M, Reiss AL; Diabetes Research in Children Network (DirecNet). Variations in Brain Volume and Growth in Young Children With Type 1 Diabetes. Diabetes. 2016 Feb;65(2):476-85. doi: 10.2337/db15-1242. Epub 2015 Oct 28. PMID 26512024
- [Background] Mauras N, Mazaika P, Buckingham B, Weinzimer S, White NH, Tsalikian E, Hershey T, Cato A, Cheng P, Kollman C, Beck RW, Ruedy K, Aye T, Fox L, Arbelaez AM, Wilson D, Tansey M, Tamborlane W, Peng D, Marzelli M, Winer KK, Reiss AL; Diabetes Research in Children Network (DirecNet). Longitudinal assessment of neuroanatomical and cognitive differences in young children with type 1 diabetes: association with hyperglycemia. Diabetes. 2015 May;64(5):1770-9. doi: 10.2337/db14-1445. Epub 2014 Dec 8. PMID 25488901
- [Background] Marzelli MJ, Mazaika PK, Barnea-Goraly N, Hershey T, Tsalikian E, Tamborlane W, Mauras N, White NH, Buckingham B, Beck RW, Ruedy KJ, Kollman C, Cheng P, Reiss AL; Diabetes Research in Children Network (DirecNet). Neuroanatomical correlates of dysglycemia in young children with type 1 diabetes. Diabetes. 2014 Jan;63(1):343-53. doi: 10.2337/db13-0179. Epub 2013 Oct 29. PMID 24170697
- [Background] Bruehl H, Sweat V, Tirsi A, Shah B, Convit A. Obese Adolescents with Type 2 Diabetes Mellitus Have Hippocampal and Frontal Lobe Volume Reductions. Neurosci Med. 2011 Mar 1;2(1):34-42. doi: 10.4236/nm.2011.21005. PMID 21691448
- [Background] Yau PL, Javier DC, Ryan CM, Tsui WH, Ardekani BA, Ten S, Convit A. Preliminary evidence for brain complications in obese adolescents with type 2 diabetes mellitus. Diabetologia. 2010 Nov;53(11):2298-306. doi: 10.1007/s00125-010-1857-y. Epub 2010 Jul 30. PMID 20668831
- [Background] Yau PL, Kang EH, Javier DC, Convit A. Preliminary evidence of cognitive and brain abnormalities in uncomplicated adolescent obesity. Obesity (Silver Spring). 2014 Aug;22(8):1865-71. doi: 10.1002/oby.20801. Epub 2014 May 28. PMID 24891029
- [Background] Cui Y, Jiao Y, Chen YC, Wang K, Gao B, Wen S, Ju S, Teng GJ. Altered spontaneous brain activity in type 2 diabetes: a resting-state functional MRI study. Diabetes. 2014 Feb;63(2):749-60. doi: 10.2337/db13-0519. Epub 2013 Dec 18. PMID 24353185
- [Background] Marder TJ, Flores VL, Bolo NR, Hoogenboom WS, Simonson DC, Jacobson AM, Foote SE, Shenton ME, Sperling RA, Musen G. Task-induced brain activity patterns in type 2 diabetes: a potential biomarker for cognitive decline. Diabetes. 2014 Sep;63(9):3112-9. doi: 10.2337/db13-1783. Epub 2014 Apr 4. PMID 24705405